CLINICAL TRIAL: NCT01348126
Title: A Randomized, Phase IIB/III Study of Ganetespib (STA-9090) in Combination With Docetaxel Versus Docetaxel Alone in Subjects With Stage IIIb or IV Non-Small-Cell Lung Cancer
Brief Title: Study of Ganetespib (STA-9090) + Docetaxel in Advanced Non Small Cell Lung Cancer
Acronym: GALAXY
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9090-08
Record Dates: First submitted 2011-05-02; First posted 2011-05-05 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Non-small Cell Lung Cancer Stage IIIB; Non-small Cell Lung Cancer Stage IV; Non-small Cell Lung Cancer Metastatic
Keywords: Advanced non-small cell lung cancer; NSCLC; Lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single agent docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel
- Combination of ganetespib and docetaxel (Experimental)
  Interventions: Drug: Combination of ganetespib and docetaxel

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m2 administered on Day 1 of a 3-week treatment cycle by 1-hour intravenous infusion
  Arms: Single agent docetaxel
Drug: Combination of ganetespib and docetaxel — Ganetespib 150 mg/m2 in combination with docetaxel 75 mg/m2. On Day 1 of each 3-week treatment cycle, ganetespib and docetaxel will be administered as separate 1-hour intravenous infusions. Ganetespib 150 mg/m2 will be administered again on Day 15 of each cycle.
  Arms: Combination of ganetespib and docetaxel

SUMMARY:
The purpose of this study is to determine whether combining ganetespib (STA-9090) with docetaxel is more effective than docetaxel alone in the treatment of subjects with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
Preliminary signals of clinical activity of ganetespib as a single agent have been observed in NSCLC. A novel approach to treatment of NSCLC is the combination of Hsp90 inhibitors, such as ganetespib, and taxanes. Such combinations have shown potential for synergy in preclinical and clinical evaluations with other Hsp90 inhibitors. Preclinical studies with ganetespib and taxanes have indicated that the combination of these drugs was more effective than either drug alone at inducing cell death, and an ongoing phase 1 study indicates that the combination is well tolerated and warrants systematic evaluation in a larger study.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of NSCLC
* Stage IIIB or IV NSCLC
* ECOG Performance Status 0 or 1
* Prior therapy defined as 1 prior systemic therapy for advanced disease
* measurable disease
* Radiologic evidence of disease progression following most recent prior treatment.
* Adequate hematologic, hepatic, renal function

Exclusion Criteria:

* Active or untreated CNS metastases
* Active malignancies other than NSCLC within the last 5 years with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri or basal or squamous cell carcinoma of the skin
* Serious cardiac illness or medical conditions
* Pregnant or lactating women
* Uncontrolled intercurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2011-05; Primary Completion 2014-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Progression-free survival in two co-primary populations | 14 months

SECONDARY OUTCOMES:
Overall Response Rate | 14 months
  ORR is the proportion of subjects who achieve tumor response
Determine qualitative and quantitative toxicities | 14 months
  AEs will be graded by NCI-CTC criteria. Tabulations of adverse events by frequency, relatedness and severity will be presented. Data will be presented by treatment arm and overall. No formal statistical analyses are planned.
Determine plasma drug concentrations of the combination | 14 months
  Assessed via measurement of Cmax levels.
Evaluate Quality of Life | 14 months
  As measured by the EORTC QLQ -C30 questionnaire
Disease Control Rate | 14 months
  Disease Control Rate is defined as the proportion of patients with best response, according to modified RECIST 1.1, of CR, PR or SD, where the SD must be for at least 6 weeks or 12 weeks.
Tumor size change | 14 months
  Tumor size changes from baseline to at least 6 and 12 weeks
Overall survival | 21 months

CONTACTS AND LOCATIONS:
Locations (49):
- United States (8):
  - Synta Pharmaceuticals Investigative Site, Tucson, Arizona
  - Synta Pharmaceuticals Investigative Site, Santa Monica, California
  - Synta Pharmaceuticals Investigative Site, Atlanta, Georgia
  - Synta Pharmaceuticals Investigative Site, Chicago, Illinois
  - Synta Pharmaceutials Investigative Site, Boston, Massachusetts
  - Synta Pharmaceuticals Investigative Site, Winston-Salem, North Carolina
  - Synta Pharmaceuticals Investigative Site, Kettering, Ohio
  - Synta Pharmaceuticals Investigative Site, Portland, Oregon
- Belgium (3):
  - Synta Pharmaceuticals Investigative Site, Brussels
  - Synta Pharmaceuticals Investigative Site, Jette
  - Synta Pharmaceuticals Investigative Site, Yvoir
- Bosnia and Herzegovina (5):
  - Synta Pharmaceuticals Investigative Site, Banja Luka
  - Synta Pharmaceuticals Investigative Site, Mostar
  - Synta Pharmaceuticals Investgative Site, Sarajevo
  - Synta Pharmaceuticals Investigative Site, Sarajevo
  - Synta Pharmaceuticals Investigative Site, Tuzla
- Canada (3):
  - Synta Pharmaceuticals Investigative Site, Hamilton
  - Synta Pharmaceuticals Investigative Site, Montreal
  - Synta Pharmaceuticals Investigative Site, Ottawa
- Croatia (3):
  - Synta Pharmaceuticals Investigative Site, Pula
  - Synta Pharmaceuticals Investigative Site, Split
  - Synta Pharmaceuticals Investigative Site, Zagreb
- Synta Pharmaceuticals Investigative Site, Prague, Czechia
- Germany (5):
  - Synta Pharmaceuticals Investigative Site, Halle
  - Synta Pharmaceuticals Investigative Site, Hamburg
  - Synta Pharmaceuticals Investigative Site, Mainz
  - Synta Pharmaceuticals Investigative Site, Mannheim
  - Synta Pharmaceuticals Investigative Site, Offenbach
- Poland (4):
  - Synta Pharmaceuticals Investigative Site, Krakow
  - Synta Pharmaceuticals Investigative Site, Olsztyn
  - Synta Pharmaceuticals Investigative Site, Prabuty
  - Synta Pharmaceuticals Investigative Site, Szczecin
- Romania (3):
  - Synta Pharmaceuticals Investigative Site, Cluj-Napoca
  - Synta Pharmaceuticals Investigative Site, Craiova
  - Synta Pharmaceuticals Investigative Site, Suceava
- Russia (5):
  - Synta Pharmaceuticals Investigative Site, Kazan'
  - Synta Pharmaceuticals Investigative Site, Moscow
  - Synta Pharmaceuticals Investigative Site, Saint Petersburg
  - Synta Pharmaceuticals Investigative Site, Sochi
  - Synta Pharmaceuticals Investigative Site, Voronezh
- Serbia (2):
  - Synta Pharmaceuticals Investigative Site, Belgrade
  - Synta Pharmaceuticals Investigative Site, Kamenitz
- Spain (3):
  - Synta Pharmaceuticals Investigative Site, Badalona
  - Synta Pharmaceuticals Investigative Site, Barcelona
  - Synta Pharmaceuticals Investigative Site, Madrid
- United Kingdom (4):
  - Synta Pharmaceuticals Investigational Site, Leicester
  - Synta Pharmaceuticals Investigative Site, London
  - Synta Pharmaceuticals Investigational Site, London
  - Synta Pharmaceuticals Investigational Site, Sutton